CLINICAL TRIAL: NCT03976271
Title: Consequences of Hypoglycaemia on Cardiovascular and Inflammatory Responses in Patients With Diabetes Mellitus Type 1, Type 2 and Healthy Volunteers
Brief Title: Consequences of Hypoglycaemia on Cardiovascular and Inflammatory Responses
Acronym: HCIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HCIR
Record Dates: First submitted 2018-11-08; First posted 2019-06-06 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-03

CONDITIONS: Hypoglycemia; Inflammatory Response; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: All subjects will undergo a hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp (nadir 2.8 mmol/L), during and after which blood and urine will be sampled for further examination for up to one week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- T1DM poor glycaemic control (Active Comparator): patients with type 1 diabetes and poor glycaemic control (HbA1c >8% / >64 mmol/mol will undergo hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
  Interventions: Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
- T1DM impaired awareness (Active Comparator): patients with type 1 diabetes and impaired awareness of hypoglycaemia will undergo hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
  Interventions: Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
- T1DM Normal awareness (Active Comparator): patients with type 1 diabetes and normal awareness of hypoglycaemia will undergo hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
  Interventions: Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
- T2DM + Insulin (Active Comparator): patients with type 2 diabetes with insulin treatment for at least 1 year will undergo hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
  Interventions: Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
- Healthy control T2DM (Active Comparator): healthy controls without diabetes and age, gender and BMI matched with diabetes type 2 participants will undergo hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
  Interventions: Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
- Healthy control T1DM (Active Comparator): Healthy controls without diabetes and age, gender and BMI matched with diabetes type 1 participants will undergo hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp
  Interventions: Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp

INTERVENTIONS:
Procedure: hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp — For this study, a hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp will be conducted to investigate the effect of hypoglycaemia. This means that subjects will receive an intravenous insulin infusion, at a continuous rate of 60 mU∙m-2∙min-1, as well as glucose 20% w/w intravenously at a variable rate, adjusted by arterial plasma glucose levels, measured at 5 minute intervals.
  Other Names: hypoglycaemic clamp

SUMMARY:
People with Type 1 diabetes (T1DM), type 2 diabetes (T2DM) and healthy volunteers will undergo a hypoglycaemic clamp to to investigate the effect of hypoglycaemia on cardiovascular and inflammatory responses.

DETAILED DESCRIPTION:
Objectives: The overall aim of the present study is to investigate the effect of hypoglycaemia on cardiovascular and inflammatory responses, molecular mechanisms and epigenetic profiles in various groups of people with diabetes type 1, type 2 and healthy volunteers.

Study design: Intervention study

Intervention: All subjects will undergo a hyperinsulinemic normoglycaemic-hypoglycaemic glucose clamp (nadir 2.8 mmol/L), during and after which blood and urine will be sampled for further examination for up to one week.

ELIGIBILITY:
Inclusion Criteria:

Overall inclusion criteria

* Ability to provide written informed consent
* Must be able to speak and read Danish (for Hillerød-site) and Dutch (for Nijmegen-site)
* Insulin treatment according to basal-bolus insulin regimen (injections or insulin pump) (except for group 5)
* Body-Mass Index: 19-40 kg/m2
* Age ≥18 years, ≤ 80 years
* Blood pressure: <140/90 mmHg
* Duration of diabetes > 1 year (except for group 5)
* HbA1c < 100 mmol/mol

Group specific

* Group 1: HbA1c >64 mmol/mol
* Group 2: impaired awareness of hypoglycaemia (IAH) as assessed by a score of ≥3 on the modified Clarke questionnaire, ≥4 on the Gold questionnaire and a positive score on the Pedersen-Bjergaard questionnaire.
* Group 3: normal awareness of hypoglycaemia (NAH) as assessed by a score of <3 on the modified Clarke questionnaire, <4 on the Gold questionnaire and a negative score on the Pedersen-Bjergaard.
* Group 4: Insulin treatment for at least 1 year
* Group 5/6: HbA1c <42 mmol/mol

Exclusion Criteria:

* - Severe medical or psychological conditions interfering with the perception of hypoglycaemia other than IAH such as brain injuries, epilepsy, a major cardiovascular disease event or anxiety disorders
* Use of immune-modifying drugs or antibiotics
* Treatment with glucose-modifying (other than insulin, SGLT-2 inhibitors and metformin) agents (e.g. prednisolon)
* Use of anti-depressive drugs
* Pregnancy or breastfeeding or unwillingness to undertake measures for birth control
* Use of statins (e.g. stop statins >2 weeks before performing blood sampling. This can be safely done in the context of primary prevention)
* Any event of cardiovascular disease in the past 5 years (e.g. myocardial infarction, stroke, heart failure, symptomatic peripheral arterial disease)
* Auto-inflammatory or auto-immune diseases
* Any infection in past three months
* Previous vaccination in the past three months
* Laser coagulation for proliferative retinopathy in the past six months
* Proliferative retinopathy
* Diabetic nephropathy as reflected by an albumin-creatinine ratio ˃ 30 mg/gor an estimated glomerular filtration rate (by MDRD) ˂60ml/min/1.73m2
* History of pancreatitis (acute or chronic) or pancreatic cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory responses of hypoglycaemia by measuring the cytokine production of isolated monocytes using ELISA | 1.5 year
  Cytokine production (TNF-alfa, IL-6, IL-10 and IL-1β) of isolated and stimulated monocytes

SECONDARY OUTCOMES:
Atherogenic responses of (recurrent) hypoglycaemia using foam cell formation. | 1.5 year
  Measurement of Ox-LDL uptake by measuring intracellular apolipoproteine B
Metabolomics profile of each group | 1.5 year
  Un-targeted metabolomics and identification of metabolites based on exact mass using metabolomics library
Epigenetic modifications | 1.5 year
  Epigenetic modifications due to hypoglycaemia in the promoter regions of the pro-inflammatory cytokines in monocytes
Cardiac function responses to hypoglycaemia using echocardiography | 1.5 year
  Cardiac function responses to hypoglycaemia using echocardiography
Cognitive function responses to hypoglycaemia using cognitive function tests (TAP, PASAT) | 1.5 year
  Amount of correct answers
Oxidative stress responses using oxidative stress marker | 1.5 year
  Excretion of guanine nucleosides in urine (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan E de Galan, MD, PhD, Principal Investigator — Radboud University Medical Center; Ulrik Pedersen-Bjergaard, MD, PhD, Principal Investigator — Nordsjællands University Hospital
Locations (2):
- Nordsjællands University Hospital, Hillerød, Nordsjaelland, Denmark
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan necessary

REFERENCES:
- [Derived] Verhulst CEM, van Heck JIP, Fabricius TW, Stienstra R, Teerenstra S, McCrimmon RJ, Tack CJ, Pedersen-Bjergaard U, de Galan BE; Hypo-RESOLVE consortium. The impact of prior exposure to hypoglycaemia on the inflammatory response to a subsequent hypoglycaemic episode. Cardiovasc Diabetol. 2024 Feb 8;23(1):55. doi: 10.1186/s12933-023-02095-w. PMID 38331900
- [Derived] Verhulst CEM, van Heck JIP, Fabricius TW, Stienstra R, Teerenstra S, McCrimmon RJ, Tack CJ, Pedersen-Bjergaard U, de Galan BE; Hypo-RESOLVE consortium. Hypoglycaemia induces a sustained pro-inflammatory response in people with type 1 diabetes and healthy controls. Diabetes Obes Metab. 2023 Nov;25(11):3114-3124. doi: 10.1111/dom.15205. Epub 2023 Jul 24. PMID 37485887
- [Derived] Verhulst CEM, Fabricius TW, Nefs G, Kessels RPC, Pouwer F, Teerenstra S, Tack CJ, Broadley MM, Kristensen PL, McCrimmon RJ, Heller S, Evans ML, Pedersen-Bjergaard U, de Galan BE. Consistent Effects of Hypoglycemia on Cognitive Function in People With or Without Diabetes. Diabetes Care. 2022 Sep 1;45(9):2103-2110. doi: 10.2337/dc21-2502. PMID 35876660